CLINICAL TRIAL: NCT06014957
Title: Comparison of Hemodynamic Effect Between the Spinal Anesthesia and Saddle Block Using Levobupivacaine During Transurethral Resection of the Prostate in Cardiac Elderly Patients: A Randomized Clinical Trial
Brief Title: Comparison of Hemodynamic Effect Between the Spinal Anesthesia and Saddle Block Using Levobupivacaine During Transurethral Resection of the Prostate in Cardiac Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Omar Twaisy, Principal investigator, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: transurethral resection
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: TURP Syndrome; Spinal Anesthesia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal group (Experimental): 12.5 mg of 0.5% hyperbaric levobupivacaine (2.5 ml) was given at the level of L4-5 interspaces after the free flow confirming of the cerebrospinal fluid (CSF),immediately positioned supine with one pillow supporting the head and shoulders.
  Interventions: Drug: spinal anesthesia
- saddle block group (Experimental): 12.5 mg of 0.5% hyperbaric levobupivacaine (2.5 ml) was given at the level of L4-5 interspaces after the free flow confirming of the cerebrospinal fluid (CSF),placed in the sitting position for ten minutes and then supine with one pillow supporting the head and shoulders.
  Interventions: Drug: saddle block

INTERVENTIONS:
Drug: spinal anesthesia — 12.5 mg of 0.5% hyperbaric levobupivacaine (2.5 ml) was given at the level of L4-5 interspaces after the free flow confirming of the cerebrospinal fluid (CSF), immediately positioned supine with one pillow supporting the head and shoulders
  Arms: spinal group
Drug: saddle block — 12.5 mg of 0.5% hyperbaric levobupivacaine (2.5 ml) was given at the level of L4-5 interspaces after the free flow confirming of the cerebrospinal fluid (CSF), placed in the sitting position for ten minutes and then supine with one pillow supporting the head and shoulders
  Arms: saddle block group

SUMMARY:
Transurethral resection of the prostate (TURP) is the most common surgical intervention for patients with benign prostatic hyperplasia. TURP is mostly applied to elderly patients with hypertension and problems with breathing, circulation system, and kidney functions; therefore, it becomes very important to keep a stable anesthesia that will minimize the hemodynamic differences in these patients. General anesthesia causes more hemodynamic differences than regional anesthesia. Thus, regional anesthesia is highly preferable in TURP applications.

DETAILED DESCRIPTION:
TURP is performed by inserting a resectoscope through the urethra and resecting prostatic tissue with an electrically powered cutting-coagulating metal loop or using laser-22 vaporization energy. This can be accomplished with either a monopolar TURP (M-TURP) or bipolar TURP (B-TURP) technique. Laser energy for TURP has also been used for many years. With each technique, as much prostatic tissue as possible is resected, but the prostatic capsule is usually preserved. If the capsule is violated, large amounts of irrigation solution can be absorbed into the circulation via the periprostatic, retroperitoneal, or peritoneal space. Bleeding during TURP is not uncommon but usually controllable; hemostasis becomes difficult when large venous sinuses are opened. If the bleeding becomes uncontrollable, the procedure should be terminated as quickly as possible, and a Foley catheter should be passed into the bladder and traction applied to it. The catheter's inflated balloon exerts lateral pressure on the prostatic bed and reduces bleeding. Bleeding requiring transfusion occurs in approximately 2.5% of TURP procedures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) III,
* with Ischemic Heart Disease (history of Myocardial Ischemia,
* a history of a positive treadmill test result (Electro Cardio Graph stress test),
* use of nitroglycerin, chronic stable angina for more than two months, or an ECG with abnormal Q waves), with ejection fraction (EF) 35%-50%,

Exclusion Criteria:

* patients under 65 years,
* patients with any diseases that increase intraabdominal pressure (any intra-abdominal mass),
* general contraindications of spinal anesthesia as patient refusal, coagulation disorders, local infection at the site of the block, psychiatric illness,

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
mean arterial blood pressure | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Omar Twaisy, New Cairo, Kharga, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharyya S, Bisai S, Biswas H, Tiwary MK, Mallik S, Saha SM. Regional anesthesia in transurethral resection of prostate (TURP) surgery: A comparative study between saddle block and subarachnoid block. Saudi J Anaesth. 2015 Jul-Sep;9(3):268-71. doi: 10.4103/1658-354X.158497. PMID 26240544
- [Background] Rooke GA, Freund PR, Jacobson AF. Hemodynamic response and change in organ blood volume during spinal anesthesia in elderly men with cardiac disease. Anesth Analg. 1997 Jul;85(1):99-105. doi: 10.1097/00000539-199707000-00018. PMID 9212130
- [Background] Gulec D, Karsli B, Ertugrul F, Bigat Z, Kayacan N. Intrathecal bupivacaine or levobupivacaine: which should be used for elderly patients? J Int Med Res. 2014 Apr;42(2):376-85. doi: 10.1177/0300060513496737. Epub 2014 Mar 4. PMID 24595149